CLINICAL TRIAL: NCT06481995
Title: Early Factor XIII Replacement in Postpartum Hemorrhage: Multi-center, Randomized, Controlled, Investigator-initiated Trial
Brief Title: SWIFT - SWIss Factor XIII Trial in PPH
Acronym: SWIFT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Christian Haslinger (Other)
Collaborators: Swiss National Science Foundation, Switzerland (Unknown)
Responsible Party: Sponsor-Investigator, Christian Haslinger, Prof. Dr. med. Christian Haslinger, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC 2024 - 00374
Record Dates: First submitted 2024-05-31; First posted 2024-07-01 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Postpartum Hemorrhage; Coagulation Disorder; Coagulation Factor Deficiency; Hemorrhage; Postpartum Complication
Keywords: Postpartum hemorrhage; coagulation factor XIII
MeSH Terms: conditions — Postpartum Hemorrhage; Hemostatic Disorders; Hemorrhage | interventions — Fibrinolysin; Factor XIII

STUDY DESIGN:
Intervention Model Description: multi- center, randomized, controlled
Who Masked: Outcomes Assessor
Masking Description: The analysis of the primary outcome will be performed using blinded treatment arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fibrogammin (FXIII) (Experimental): Women in the intervention group receive FXIII intravenously in addition to the standard of care treatment for PPH. FXIII is administered when blood loss is > 700 ml. Women weighing <80 kg receive 1250 IU Fibrogammin®; women weighing 80-99.9 kg receive 1500 IU Fibrogammin®; thus ensuring a dose of 15-20 IU FXIII per kg body weight according to the manufacturer's recommendation.
  Interventions: Drug: Fibrogammin
- Control (No Intervention): Women in the control group will be treat according to the standard of care procedure for PPH.

INTERVENTIONS:
Drug: Fibrogammin — Fibrogammin is administered according to the Summary of product characteristics (SmPC) after measured blood loss exceeds 700 ml and bleeding is ongoing
  Other Names: Factor XIII
  Arms: Fibrogammin (FXIII)

SUMMARY:
The goal of this trial is to determine if postpartum blood loss can be reduced by replenishing coagulation factor XIII (FXIII) at an early stage of postpartum hemorrhage (PPH).

Summary of current body of evidence:

* Morbidity and mortality due to PPH is rising.
* Current guidelines focus on replenishment of fibrinogen as an initial step in the treatment of PPH-related coagulopathy, despite non-conclusive evidence in all prospective trials.
* Trials from other specialties demonstrate a significant impact of FXIII on perioperative bleeding complications; a previous study at the University Hospital Zurich showed that pre-partum factor XIII activity had a strong association to postpartum blood loss.

Therefore, this nationwide, multi-center, randomized, controlled trial in multiple perinatal centers across Switzerland will be conducted. The goal is to determine if postpartum blood loss and PPH-related complications can be reduced by replenishing FXIII.

All participating women receive, according to the national guideline, 1g tranexamic acid (TXA) i.v. in case of PPH (measured blood loss [MBL] ≥ 500 mL) during the pre-study phase. Randomization takes place if bleeding continues and exceeds 700mL. The intervention group then receives FXIII (Fibrogammin®) according to approved dosage in addition to obstetric standard of care treatment for causes of PPH; the control group receives only standard of care treatment.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is a main reason for maternal mortality and morbidity. PPH, defined by the WHO as blood loss of 500 mL or more within 24 hours after delivery, causes about 30% of maternal deaths worldwide. The internationally observed trend towards increased PPH-related morbidity and mortality is disturbing and demands new strategies in the prevention and treatment of PPH.

Although the most frequent causes for severe PPH are believed to be uterine atony or retained placenta, virtually all cases of severe PPH lead to a disorder of the coagulation system which itself aggravates bleeding.

At the moment, most guidelines on coagulation management during PPH and expert opinions focus on the replenishment of coagulation factor I (fibrinogen) although three out of three randomized controlled trials with early or pre-emptive administration of fibrinogen during PPH were negative.

Based on earlier research, it was hypothesized that coagulation factor XIII (FXIII) might play a significant role in women with increased postpartum blood loss, because of its role in the establishment of blood clot stability and fibrinolytic resistance. This hypothesis was tested in a prospective diagnostic study involving 1300 parturient women at the University Hospital Zurich and showed that pre-partum factor XIII activity had a strong association to postpartum blood loss.

Therefore, this nationwide, multi-center, open-label, randomized controlled trial in major perinatal centers across Switzerland will be conducted. The goal is to determine if postpartum blood loss and PPH-related complications can be reduced by substitution of FXIII at an early stage of PPH.

Irrespective of the answer to the question whether FXIII is effective in the treatment of PPH, this trial will contribute to enhancing the comprehension of coagulopathy in the context of PPH

ELIGIBILITY:
Inclusion Criteria:

* planned vaginal delivery
* singleton vital pregnancy
* gestational age at delivery >= 30+0 weeks
* maternal weight at admission for delivery <100 kg

Exclusion Criteria:

* Antithrombotic therapy in pregnancy (therapeutic dosage) until admission for delivery (LMWH, UFH)
* diagnosis of preeclampsia (ISSHP classification , eclampsia or HELLP syndrome),
* known history of deep vein thrombosis or pulmonary embolism,
* known diagnosis of bleeding disorder or thrombophilia,
* known thrombocytopenia during second half of pregnancy with thrombocytes < 100 G/L,
* known anemia during second half of pregnancy with Hb<80 g/L,
* known sickle cell disease,
* known malignant tumor(s),
* participation in another study with investigational drug within the 30 days preceding and during the present study,
* inability to follow the procedures of the study, e.g. due to language problems,
* known or suspected non-compliance, drug or alcohol abuse.

Exclusion criteria prior randomization

* Maternal fever ≥39.0°C
* unplanned cesarean delivery is performed,
* Measured Blood Loss remains < 700 mL after administration of 1g tranexamic acid .
* Postpartum hemorrhage due to occult bleeding (intra-abdominal, retroperitoneal, parametric),

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 988 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Loss during post partum hemorrhage | Day 1 (within 24 hours after delivery)
  Measured blood loss, in ml

SECONDARY OUTCOMES:
Outcome of postpartum hemorrhage | Time point of assessment will be 48 hours (range 36 to 60) postpartum, if not stated otherwise
  Composite of adverse maternal outcomes related to postpartum hemorrhage, including postpartum hemorrhage with measure blood loss ≥2000 mL (within 24 hours), admission to intensive care unit, blood transfusion, need for embolization of the pelvic arteries, laparotomy with surgical measures (such as compression sutures, or ligatures), or hysterectomy during hospitalization.
Changes in hematological standard value: hemoglobin | shortly before delivery and 48 hours (range 36 to 60 hours) after delivery
  Comparison of hemoglobin values, pre-partum and post-partum (in g/L)
Changes in hematological standard value: leucocyte count | shortly before delivery and 48 hours (range 36 to 60 hours) after delivery
  Comparison of leucocyte count, pre-partum and post-partum (in G/l)
Changes in hematological standard value; thrombocyte count | shortly before delivery and 48 hours (range 36 to 60 hours) after delivery
  Comparison of thrombocyte count, pre-partum and post-partum (in G/l)
Hospital costs | from admission to hospital until hospital discharge, up to 9 weeks
  Total costs (in CHF)
Breastfeeding | 6 - 9 weeks after delivery
  Number of women who exclusively breastfeed their babies after PPH
Patient survey (in a subgroup of patients only) | discharge from hospital, estimated 3 - 5 days after delivery
  Questionnaire for personal experience during PPH

OTHER OUTCOMES:
Thromboembolic events | 6 - 9 weeks after delivery (visit 4)
  Number of thromboembolic events (safety outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Haslinger, Prof. Dr., Study Chair — University of Zurich; Begoña Martinez de Tejada, MD PhD, Principal Investigator — University Hospital, Geneva; David Baud, MD PhD, Principal Investigator — University of Lausanne Hospitals; Beatrice Mosimann, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland; Tina Fischer, MD, Principal Investigator — Cantonal Hospital of St. Gallen; Leonhard Schäffer, Prof. Dr., Principal Investigator — Kantonsspital Baden; Michael Winter, MD, Principal Investigator — Spital Zollikerberg; Jarmila Zdanowicz, MD, Principal Investigator — Inselspital-University Hospital Bern; Leila Sultan-Beyer, MD, Principal Investigator — Cantonal Hospital Winterthur
Locations (9):
- Switzerland (9):
  - University Hospital Geneva, Geneva, Canton of Geneva
  - Cantonal Hospital Winterthur, Winterthur, Canton of Zurich
  - Spital Zollikerberg, Zollikerberg, Canton of Zurich
  - University Hospital of Zurich, Zurich, Canton of Zurich
  - Cantonal Hospital Baden, Baden
  - University Hospital Basel, Basel
  - Inselspital-University Hospital Bern, Bern
  - University Hospital Lausanne, Lausanne
  - Cantonal Hospital St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Yes
The data sharing plan aims to ensure computational reproducibility of all published research findings obtained from data collected in this trial. Each publication will be accompanied by a dedicated compendium containing deidentified individual patient data necessary to independently reproduce the analyses presented in the corresponding publication. Such a compendium also contains information about the computer code that was used to generate figures, tables, and other statistical output. Distribution will be via a data repository following FAIR principles (such as zenodo.org).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: At the time of publication
Access Criteria: Access will be provided without limitations. Data will be provided to allow independent computational reproducibility of already published results.

REFERENCES:
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] GBD 2015 Maternal Mortality Collaborators. Global, regional, and national levels of maternal mortality, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1775-1812. doi: 10.1016/S0140-6736(16)31470-2. PMID 27733286
- [Background] Weeks A. The prevention and treatment of postpartum haemorrhage: what do we know, and where do we go to next? BJOG. 2015 Jan;122(2):202-10. doi: 10.1111/1471-0528.13098. Epub 2014 Oct 7. PMID 25289730
- [Background] WHO Recommendations for the Prevention and Treatment of Postpartum Haemorrhage. Geneva: World Health Organization; 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK131942/ PMID 23586122
- [Background] Haslinger C, Korte W, Hothorn T, Brun R, Greenberg C, Zimmermann R. The impact of prepartum factor XIII activity on postpartum blood loss. J Thromb Haemost. 2020 Jun;18(6):1310-1319. doi: 10.1111/jth.14795. Epub 2020 Apr 16. PMID 32176833
- [Background] Korte WC, Szadkowski C, Gahler A, Gabi K, Kownacki E, Eder M, Degiacomi P, Zoller N, Devay J, Lange J, Schnider T. Factor XIII substitution in surgical cancer patients at high risk for intraoperative bleeding. Anesthesiology. 2009 Feb;110(2):239-45. doi: 10.1097/ALN.0b013e318194b21e. PMID 19194150
- [Background] Wettstein P, Haeberli A, Stutz M, Rohner M, Corbetta C, Gabi K, Schnider T, Korte W. Decreased factor XIII availability for thrombin and early loss of clot firmness in patients with unexplained intraoperative bleeding. Anesth Analg. 2004 Nov;99(5):1564-1569. doi: 10.1213/01.ANE.0000134800.46276.21. PMID 15502066
- [Derived] Haslinger C, Hothorn T, Bossung V, Kalimeris S, Ranieri E, Ochsenbein-Koelble N, Korte W. Effects of early factor XIII replacement in postpartum hae morrhage: study protocol for a multicentre, open-label, randomised, controlled, investigator-initiated trial. BMJ Open. 2025 May 8;15(5):e100262. doi: 10.1136/bmjopen-2025-100262. PMID 40345697